CLINICAL TRIAL: NCT00753857
Title: The Drug Facts Box: Helping Consumers Understand Drugs for Risk Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Lisa Schwartz, VA Outcomes Group
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DMS-15879-2; NCT00386932
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: risk communication; probability sample by random digit dialing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants received 2 ads for drugs to reduce cardiovascular risk with drug facts boxes second pages.
  Interventions: Other: Drug Facts Box
- 2 (Active Comparator): Participants receive the same 2 advertisements for drugs to reduce cardiovascular risk with the standard second page (i.e., brief summary)
  Interventions: Other: Standard Brief Summary

INTERVENTIONS:
Other: Drug Facts Box — Educational intervention of 1 page summary of drug efficacy and side effects
  Arms: 1
Other: Standard Brief Summary — Ads consisted of the standard second page called the brief summary
  Arms: 2

SUMMARY:
RATIONALE:

The way in which information about a drug is provided may affect the ability of patients and doctors to understand how a drug works and the side effects of the drug.

PURPOSE:

This randomized trial is studying how well a drug facts page works compared with a short drug summary in helping patients and doctors understand medical information.

DETAILED DESCRIPTION:
This is a randomized study. Participants are contacted by phone via random-digit dialing for initial interview using the computer-assisted telephone interviewing (CATI) system. Eligible participants are then randomized to 1 of 2 intervention arms.

* Compare the effect of a prescription drug summary (one-page summary of drug information that includes a table with data on drug benefit and side effects) vs standard brief summary in direct-to-consumer advertisements on the comparisons of two drugs for the same indication, knowledge of drug efficacy and side effects of each drug, perceptions of drug efficacy and side effects of each drug
* Comprehension of information contained in the drug facts box

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70 year old in household selected by random digit dialing

Exclusion Criteria:

* Non-English speaking

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Comparison of two drugs for the same indication, Knowledge and judgments about 2 drugs to reduce the future risk of cardiovascular events | Immediate return of patient survey

SECONDARY OUTCOMES:
Comprehension of information contained in the drug facts box | Immediate return of patient survey

CONTACTS AND LOCATIONS:
Overall Officials: Steven Woloshin, MD, MS, Principal Investigator — Dartmouth Medical School; VA Medical Center (WRJ); Lisa M Schwartz, MD, MS, Principal Investigator — Dartmouth Medical School, VA Medical Center (WRJ)
Locations (1):
- VA Medical Center, White River Junction, Vermont, United States